CLINICAL TRIAL: NCT04194346
Title: Determination of Normal Values of Regional Pulmonary Strain Using a New Ultrasonographic Tool in Healthy Volunteers
Acronym: Strain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19.251
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Intervention Model Description: Prospective, interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Determination of local pleural strain (Experimental): The average Von Mises coefficient will be calculated for each recorded ultrasound loop using a non-invasive vascular elastography platform.
  Interventions: Procedure: Lung ultrasound

INTERVENTIONS:
Procedure: Lung ultrasound — Healthy volunteers will have lung ultrasonography at 15 predetermined sites for a common volume continuum between 5 and 15 cc/kg. For each volume, 3 respiratory cycles will be recorded.

SUMMARY:
Mechanical ventilation is frequently used in the operating room and the intensive care settings. Although essential in many cases, mechanical ventilation can be responsible for ventilator-induced lung injury (VILI). The relationship between mechanical ventilation and VILI has been clearly demonstrated in animals and is highly suspected in humans. The putative mechanism responsible for VILI is excessive pulmonary strain or overdistension. Frequently observed in mechanically ventilated patients, the presence of a severe pre-existing pulmonary disease can increase the risk of overdistension. The development of a tool allowing early detection of pulmonary overdistension would represent a great asset in the prevention of VILI by allowing safer adjustments of mechanical ventilation parameters. Ultrasonographic imaging is a non-radiant, non-invasive technique already available in the intensive care setting. Already used for cardiac strain measurements, ultrasonography is a promising avenue to assess pulmonary strain.This study will aim to establish normal pleural strain values using ultrasonography in healthy volunteers.

Purpose: The primary objective is to calculate 95% confidence intervals in pleural strain for a set of 8 inspired volumes at 15 predetermined lung areas in healthy volunteers.

The secondary objectives of the study are:

* to modelize the relation between pleural strain and inspired volume
* to modelize the relation between pleural strain and global pulmonary volumetric strain
* to modelize the relation between pleural strain and maximal echo intensity change
* to compare the regional distribution pattern of pleural strain in healthy volunteers in dependent versus non-dependent areas.

Hypothesis: Elastography using the Lagrangian speckle model estimator based on optical flow allows the determination of normal mean values and 95% confidence intervals of pleural strain (average Von Mises coefficient) in 15 predetermined lung areas for a set of 8 inspired volumes in healthy volunteers.

DETAILED DESCRIPTION:
Participants will have their functional residual capacity (FRC) measured by a nitrogen dilution technique. Subsequently, they will be instructed to breathe 8 different inspired volumes (5 to 15 ml/kg predicted body weight). Tidal volumes will be measured using a spirometer. For each inspired volume, 3 respiratory cycles will be recorded at 15 predetermined anatomic sites: 1st and 3rd left and right intercostal spaces at the mid-clavicular line, 5th right intercostal space at the mid-clavicular line, 2nd, 4th and 6th left and right intercostal spaces at the anterior axillary line, and 5th and 7th left intercostal spaces and right to the posterior axillary line. For each image, the probe will be oriented perpendicularly to the ribs. A research, non-commercially available, non-invasive vascular elastography platform will be used to calculate the various strain parameters for all of the recorded cineloops. For each recorded clip, an experienced lung ultrasonographer will segment the pleura on a single reference image. From this image, an algorithm will define a region of interest which will be tracked throughout the rest of the images of the video sequence. Finally, the algorithm will calculate the various components of pleural strain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (20 men/20 women)
* 18 years old and over
* Functional capacity superior to 4 METs (metabolic equivalent of task)

Exclusion Criteria:

* Previous thoracic procedure (chest tube, thoracotomy, thoracoscopy)
* Pre-existing pulmonary disease (asthma, chronic obstructive pulmonary disease, lung fibrosis)
* Active or previous history of smoking
* Obesity (Body Mass Index superior to 30 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — An equal number of men and women will be recruited.
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Average Von Mises | At the end of the study on Day 1
  Three respiratory cycles will be analyzed using an elastography technique based on optical flow to calculate the average Von Mises coefficient. The mean value will be retained.

SECONDARY OUTCOMES:
Sum of the ranges of cumulated absolute axial and cumulated absolute lateral deformation | At the end of the study on Day 1
  Three respiratory cycles will be analyzed using an elastography technique based on optical flow to calculate the sum of the ranges of cumulated absolute axial and cumulated absolute lateral deformation in percentage for each cycle. The mean value will be retained.
Range of cumulated absolute lateral deformation | At the end of the study on Day 1
  Three respiratory cycles will be analyzed using an elastography technique based on optical flow to calculate the range of cumulated absolute lateral deformation in percentage for each respiratory cycle. The mean value will be retained.
Cumulated absolute lateral translation | At the end of the study on Day 1
  Three respiratory cycles will be analyzed using an elastography technique based on optical flow to calculate the cumulated absolute lateral translation in millimeters for each respiratory cycle. The mean value will be retained.
Maximal echo intensity change | At the end of the study on Day 1
  Three respiratory cycles will be analyzed to calculate the maximal echo intensity change using an ordinal scale from 0 to 255. The mean value will be retained.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No